CLINICAL TRIAL: NCT04435327
Title: SequelaeCov: a Prospective Study on Lung Damage Caused by SARS-CoV-2 Pneumonia
Brief Title: Lung Damage Caused by SARS-CoV-2 Pneumonia (COVID-19)
Acronym: SequelaeCov
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: SequelaeCov
Record Dates: First submitted 2020-06-12; First posted 2020-06-17 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-01

CONDITIONS: COVID; Pneumonia, Viral; Barotrauma; Interstitial Lung Disease; Bronchiectasis Adult; Emphysema
MeSH Terms: conditions — Pneumonia, Viral; Barotrauma; Lung Diseases, Interstitial; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Oxygen therapy: Patients who were hospitalised due to COVID-19 pneumonia and received only oxygen support therapy.
- Non invasive ventilation (NIV/CPAP): Patients who were hospitalised due to COVID-19 pneumonia and received non invasive ventilation (NIV/CPAP) as maximum support therapy
- Invasive ventilation: Patients who were hospitalised due to COVID-19 pneumonia and received invasive mechanical ventilation (IMV)

SUMMARY:
Pneumonia is a recurrent element of COVID-19 infection, it is often associated with development of respiratory failure and patients frequently need various degrees of oxygen therapy up to non invasive ventilation (NIV-CPAP) and invasive mechanical ventilation (IMV).

Main purpose of this study is to evaluate with non invasive clinical instruments (pletysmography, Diffusion lung capacity for carbon monoxide -DLCO-, six minute walking test and dyspnea scores) and radiological tools (chest X-ray and chest CT scan) the development of medium-to-long term pulmonary sequelae caused by SARS-CoV-2 pneumonia.

DETAILED DESCRIPTION:
SARS-CoV-2 related disease started in December 2019 in the Chinese city of Wuhan, rapidly spread and became an international health emergency.

Pneumonia is a frequent element of COVID-19, its pathogenic mechanisms are not entirely known and some patients develop various degrees of respiratory failure and need oxygen therapy up to NIV-CPAP) and IMV.

Some pathology studies in COVID-19 pneumonia show ARDS-like lesions associated to inflammatory reaction. It is known that pulmonary inflammatory damage can lead to fibrotic sequelae or to the development of pulmonary emphysema.

The main target of the study is to use non invasive methods (pletysmography, DLCO assessment, six minute walking test and dyspnea scores) and radiological tools (chest X-ray and chest CT scan) to identify pulmonary sequelae in patients hospitalised because of respiratory failure in COVID-19 pneumonia.

Study design: multicentre observational cohort study. Patients will be divided in three arms according to maximum ventilatory/oxygen support received during hospital stay:

1. patients who received only oxygen therapy
2. patients who received non invasive ventilation (NIV-CPAP)
3. patients who received invasive mechanical ventilation (IMV)

All patients undergo a clinical evaluation at 6 months from hospital discharge (T1) and a second clinical evaluation at 12 months from hospital discharge (T2).

During (T1) patients undergo spirometry with pletysmography and DLCO assessment, six minute walking test, standard chest X-ray, arterial blood gas analysis if SaO2 < 93% in room air, dyspnea score and presence and extension of lung sounds at pulmonary auscultation.

During (T2) patients will undergo spirometry with pletysmography and DLCO assessment, six minute walking test, High Resolution CT scan (HRTC) of the thorax, arterial blood gas analysis if SaO2 < 93% in room air, dyspnea score and presence and extension of lung sounds at pulmonary auscultation).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years
* Able to sign informed consent to participate in the study
* Real time PCR diagnosis od SARS-CoV-2 infection
* Hospital admission due to clinical/instrumental diagnosis of interstitial pneumonia
* Presence of acute respiratory failure (PaO2/FiO2 <300 mm Hg) at the moment of hospital admission

Exclusion Criteria:

* Severe renal failure defined as glomerular filtration rate (GFR) < 30 ml/min at hospital discharge
* Cardiovascular failure NYHA class IV (patient unable to perform any activity) at hospital discharge
* Active solid or hematological malignancies at hospital discharge
* Prior diagnosis of chronic obstructive pulmonary disease (COPD), pulmonary emphysema, pulmonary fibrosis, bronchiectasis associated or not associated to cystic fibrosis
* Pregnancy or breastfeeding
* Suspected bacterial or fungine pulmonary superinfection during hospital stay

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with respiratory failure (P/F < 300) due to SARS-CoV-2 pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Reduction of Diffusion of Lung CO (DLCO, single breath technique) | T1 at 6 months from discharge
  Reduction below 80% of predicted values of DLCO
Reduction of Diffusion of Lung CO (DLCO, single breath technique) | T2 at 12 months from discharge
  Reduction below 80% of predicted values of DLCO

SECONDARY OUTCOMES:
Alterations in 6 minute walking test (6MWT) | T1 at 6 months from discharge
  reduction in maximum distance walked
Alterations in 6 minute walking test (6MWT) | T2 at 12 months from discharge
  reduction in maximum distance walked
Alterations in 6 minute walking test (6MWT) | T1 at 6 months from discharge
  reduction in oxygen saturation nadir
Alterations in 6 minute walking test (6MWT) | T2 at 12 months from discharge
  reduction in oxygen saturation nadir
Alterations of pletismography | T1 at 6 months from discharge
  reduction of Forced Vital Capacity (FVC, %)
Alterations of pletismography | T2 at 12 months from discharge
  reduction of Forced Vital Capacity (FVC, %)
Alterations of pletismography | T1 at 6 months from discharge
  reduction of Forced Vital Capacity (FVC, L)
Alterations of pletismography | T2 at 12 months from discharge
  reduction of Forced Vital Capacity (FVC, L)
Alterations of pletismography | T1 at 6 months from discharge
  reduction of Vital Capacity (VC, %)
Alterations of pletismography | T2 at 12 months from discharge
  reduction of Vital Capacity (VC, %)
Alterations of pletismography | T1 at 6 months from discharge
  reduction of Vital Capacity (VC, L)
Alterations of pletismography | T2 at 12 months from discharge
  reduction of Vital Capacity (VC, L)
Alterations of pletismography | T1 at 6 months from discharge
  reduction of Forced Expiratory Volume in the 1st second (FEV1, L)
Alterations of pletismography | T1 at 6 months from discharge
  reduction of Forced Expiratory Volume in the 1st second (FEV1, %)
Alterations of pletismography | T2 at 12 months from discharge
  reduction of Forced Expiratory Volume in the 1st second (FEV1, L)
Alterations of pletismography | T2 at 12 months from discharge
  reduction of Forced Expiratory Volume in the 1st second (FEV1, L%)
Alterations of pletismography | T1 at 6 months from discharge
  reduction of Total Lung Capacity (TLC, L)
Alterations of pletismography | T1 at 6 months from discharge
  reduction of Total Lung Capacity (TLC, %)
Alterations of pletismography | T2 at 12 months from discharge
  reduction of Total Lung Capacity (TLC, L)
Alterations of pletismography | T2 at 12 months from discharge
  reduction of Total Lung Capacity (TLC, %)
Alterations of pletismography | T1 at 6 months from discharge
  alterations of Residual Volume (RV,%)
Alterations of pletismography | T1 at 6 months from discharge
  alterations of Residual Volume (RV, L)
Alterations of pletismography | T2 at 12 months from discharge
  alterations of Residual Volume (RV, L)
Alterations of pletismography | T2 at 12 months from discharge
  alterations of Residual Volume (RV, %)
Alterations of pletismography | T1 at 6 months from discharge
  increase of Specific Airway Resistance (sRAW) (absolute value)
Alterations of pletismography | T1 at 6 months from discharge
  increase of Specific Airway Resistance (sRAW) (%)
Alterations of pletismography | T2 at 12 months from discharge
  increase of Specific Airway Resistance (sRAW) (absolute value)
Alterations of pletismography | T2 at 12 months from discharge
  increase of Specific Airway Resistance (sRAW) (%)
Alterations of pletismography | T1 at 6 months from discharge
  alterations of Motley Index (VR/CPT)
Alterations of pletismography | T2 at 12 months from discharge
  alterations of Motley Index (VR/CPT)
Alterations of pletismography | T1 at 6 months from discharge
  alterations of Tiffeneau Index (IT)
Alterations of pletismography | T2 at 12 months from discharge
  alterations of Tiffeneau Index (IT)
Alterations of Arterial Blood Gas Analysis | T1 at 6 months from discharge
  reduction of PaO2 mmHg
Alterations of Arterial Blood Gas Analysis | T2 at 12 months from discharge
  reduction of PaO2 mmHg
Alterations of Arterial Blood Gas Analysis | T1 at 6 months from discharge
  alteration of PaCO2 mmHg
Alterations of Arterial Blood Gas Analysis | T2 at 12 months from discharge
  alteration of PaCO2 mmHg
Abnormal Dyspnea Score | T1 at 6 months from discharge
  Modified Medical Research Council - mMRC > 0 (minimum 0, maximum 4; higher score means worse outcome)
Abnormal Dyspnea Score | T2 at 12 months from discharge
  Modified Medical Research Council - mMRC > 0(minimum 0, maximum 4; higher score means worse outcome)
Presence and extension of abnormal pulmonary lung sounds at auscultation | T1 at 6 months from discharge
  Presence and extension of abnormal pulmonary lung sounds at auscultation
Presence and extension of abnormal pulmonary lung sounds at auscultation | T2 at 12 months from discharge
  Presence and extension of abnormal pulmonary lung sounds at auscultation
Presence and extension of radiological alterations at chest X-ray | T1 at 6 months from discharge
  Presence and extension of radiological alterations at chest X-ray
Presence and extension of radiological alterations at chest CT scan | T2 at 12 months from discharge
  Presence and extension of radiological alterations at chest CT scan

CONTACTS AND LOCATIONS:
Locations (1):
- San Gerardo Hospital, Monza, MB, Italy

REFERENCES:
- [Result] Faverio P, Luppi F, Rebora P, Busnelli S, Stainer A, Catalano M, Parachini L, Monzani A, Galimberti S, Bini F, Bodini BD, Betti M, De Giacomi F, Scarpazza P, Oggionni E, Scartabellati A, Bilucaglia L, Ceruti P, Modina D, Harari S, Caminati A, Valsecchi MG, Bellani G, Foti G, Pesci A. Six-Month Pulmonary Impairment after Severe COVID-19: A Prospective, Multicentre Follow-Up Study. Respiration. 2021;100(11):1078-1087. doi: 10.1159/000518141. Epub 2021 Aug 19. PMID 34515212